CLINICAL TRIAL: NCT07058948
Title: A Phase II Prospective, Open-Label, Single-Arm Study Evaluating the Efficacy and Safety of Spatially Fractionated Radiotherapy Combined With Immunotherapy in Patients With Advanced Solid Tumors
Brief Title: Spatially Fractionated Radiotherapy Combined With Immunotherapy for Advanced Solid Tumors
Acronym: SFRT-IM-P2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20250717
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Solid Cancers; Radiotherapy; Immune Checkpoint Inhibitor; Lung Cancer
Keywords: spatially fractionated radiotherapy; solid cancers; immune checkpoint inhibitor
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Eligible patients in this Phase II trial will undergo specific - dose irradiation using a medical linear accelerator. Within the largest tumor's gross tumor volume (GTV), spheres (0.5 - 3 cm in diameter) will be created as high - dose targets (LRT targets), spaced 2.0 - 5.0 cm apart. The LRT targets must be drawn within the GTV, avoiding blood vessels, with a margin of at least 1 cm from the GTV edge and a volume ratio of 1% - 10% of the GTV.
  For a single lesion, the D95 of the GTV will be ≥1 Gy per fraction, and the D95 of the LRT target will be 8 - 12 Gy per fraction, while keeping the single - fraction dose to organs at risk as low as possible. All other irradiated metastases will receive low - dose radiotherapy at 100 - 300 cGy × 5 fractions. Brain and bone metastases will be treated with palliative radiotherapy as per clinical routine and are not included in the low - dose radiotherapy. Immunotherapy will be administered during or within one week after radiotherapy.
  Interventions: Radiation: lattice radiation therapy

INTERVENTIONS:
Radiation: lattice radiation therapy — Eligible patients will receive treatment using a medical linear accelerator. Within the largest tumor's gross tumor volume (GTV), spheres (0.5 - 3 cm in diameter) will be created as high - dose targets (LRT targets), spaced 2.0 - 5.0 cm apart. The LRT targets must be drawn within the GTV, avoiding blood vessels, with a margin of at least 1 cm from the GTV edge and a volume ratio of 1% - 10% of the GTV.
  For a single lesion, the D95 of the GTV will be ≥1 Gy per fraction, and the D95 of the LRT target will be 8 - 12 Gy per fraction, while keeping the single - fraction dose to organs at risk as low as possible. All other irradiated metastases will receive low - dose radiotherapy at 100 - 300 cGy × 5 fractions. Brain and bone metastases will be treated with palliative radiotherapy as per clinical routine and are not included in the low - dose radiotherapy. Immunotherapy will be administered during or within one week after radiotherapy.

SUMMARY:
Lattice radiation therapy (LRT) is a spatially fractionated radiotherapy technique that creates alternating high - and low - dose areas within a tumor to enhance local control and reduce toxicity to surrounding tissues. This study aims to evaluate the effectiveness and safety of combining LRT with immunotherapy in patients with advanced or metastatic solid tumors, through a Phase II clinical trial. Patients will receive specific - dose irradiation using a medical linear accelerator. Within the GTV of the largest tumor, spheres (0.5 - 3 cm in diameter) will be created as high - dose targets (LRT targets), spaced 2.0 - 5.0 cm apart. The LRT targets must be drawn within the GTV, avoiding blood vessels, with a margin of at least 1 cm from the GTV margin, and a volume ratio of 1% - 10% of the GTV. For a single lesion, the D95 of the GTV will be ≥1 Gy/fraction, and the D95 of the LRT target will be 8 - 12 Gy/fraction, with minimal possible single - fraction doses to organs at risk. All other irradiated metastases will receive low - dose radiotherapy (100 - 300 cGy × 5 fractions), except for brain and bone metastases, which will be treated with palliative radiotherapy as per clinical routine. Immunotherapy will be administered during or within one week after radiotherapy.

DETAILED DESCRIPTION:
This Phase II clinical trial investigates the combination of lattice radiation therapy (LRT) and immunotherapy in patients with advanced or metastatic solid tumors. LRT, a spatially fractionated radiotherapy technique, creates alternating high - and low - dose regions within the tumor to enhance local control and reduce toxicity to surrounding tissues.

Eligible patients will receive treatment using a medical linear accelerator. Within the largest tumor's gross tumor volume (GTV), spheres (0.5 - 3 cm in diameter) will be created as high - dose targets (LRT targets), spaced 2.0 - 5.0 cm apart. The LRT targets must be drawn within the GTV, avoiding blood vessels, with a margin of at least 1 cm from the GTV edge and a volume ratio of 1% - 10% of the GTV.

For a single lesion, the D95 of the GTV will be ≥1 Gy per fraction, and the D95 of the LRT target will be 8 - 12 Gy per fraction, while keeping the single - fraction dose to organs at risk as low as possible. All other irradiated metastases will receive low - dose radiotherapy at 100 - 300 cGy × 5 fractions. Brain and bone metastases will be treated with palliative radiotherapy as per clinical routine and are not included in the low - dose radiotherapy. Immunotherapy will be administered during or within one week after radiotherapy.

The study will monitor patients for treatment - related toxicities, immune - related adverse events, and assess treatment efficacy through imaging studies and biomarker analysis. The results will provide insights into the effectiveness and safety of combining LRT with immunotherapy for advanced solid tumors.

ELIGIBILITY:
**Inclusion Criteria:**

1. Signed informed consent.
2. Histologically or cytologically confirmed malignant solid tumor.
3. Advanced solid tumor unsuitable for surgery as determined by a multidisciplinary tumor board or consulting physicians.
4. No available standard therapy or inability to tolerate it, with imaging and clinical assessment showing stable disease (SD) or progressive disease (PD).
5. Age ≥18 years on the day of signing informed consent.
6. No prior radiotherapy to the proposed site, or last radiotherapy ≥6 months ago.
7. KPS score ≥70.
8. At least one measurable lesion per RECIST 1.1. Previously irradiated lesions qualify only if significant progression post - radiotherapy.
9. Life expectancy >3 months.
10. Adequate organ and bone marrow function:

    * Marrow: ANC ≥1.5×10⁹/L, platelets ≥80×10⁹/L, hemoglobin ≥9 g/dL;
    * Liver: Total bilirubin ≤1.5× upper limit of normal (ULN), ALT/AST ≤1.5× ULN;
    * Kidney: Serum creatinine ≤1.5× ULN or creatinine clearance ≥50 ml/min, blood urea nitrogen ≤200 mg/L;
    * Coagulation: INR ≤1.5× ULN, PTT ≤1.5× ULN.
11. Recovery from prior therapy - related adverse events (≤Grade 1 or baseline).
12. Willingness to use appropriate contraception.
13. No radiotherapy contraindications as judged by the radiation oncologist.
14. Agreement to receive both immunotherapy and radiotherapy.

**Exclusion Criteria:**

1. Active central nervous system (CNS) metastases, carcinomatous meningitis, or spinal cord compression.
2. Severe comorbidities such as myocardial infarction within 6 months, severe arrhythmias, or psychosis that may affect treatment completion or result in a life expectancy of <3 months.
3. Evidence of interstitial lung disease or active/non - infectious pneumonia (e.g., drug - induced, radiation - induced) requiring steroid treatment.
4. History of pulmonary fibrosis, pulmonary artery hypertension, or severe irreversible airway obstruction.
5. Presence of peripheral neuropathy.
6. Severe organ dysfunction (e.g., hepatic, cardiopulmonary failure) that is likely to make radiotherapy intolerable.
7. Known allergy to study drugs or excipients, or a history of severe allergic reaction to any PD - 1 monoclonal antibody.
8. Serious infection within 4 weeks prior to the start of study treatment, including but not limited to hospitalization for infection, bacteremia, or severe pneumonia; or receipt of oral or intravenous antibiotics within 2 weeks prior to study treatment. Patients receiving prophylactic antibiotics (e.g., for urinary tract infections or chronic obstructive pulmonary disease exacerbations) are eligible.
9. Known or suspected active autoimmune disease (e.g., uveitis, colitis, hepatitis, hypophysitis, vasculitis, nephritis, thyroiditis). Exceptions: patients with vitiligo, cured childhood asthma; patients with well - controlled type 1 diabetes on insulin.
10. History of allogeneic organ transplant (except corneal) or allogeneic hematopoietic stem cell transplant.
11. Pregnant or breastfeeding women.
12. Any other condition that the investigator deems a valid reason for disqualification based on the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Assessed at 6 weeks post-treatment initiation
  The primary endpoint is the objective response rate, measuring tumor reduction usingRECIST v1.1 criteria.

SECONDARY OUTCOMES:
Adverse Events | During and up to 1year post - treatment.
  Incidence and grading of Adverse Events (AEs) and Serious Adverse Events (SAEs) (assessed using the NCI CTCAE v5.0 criteria), including abnormalities in vital signs, electrocardiograms, and laboratory tests

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No